CLINICAL TRIAL: NCT04431713
Title: An Open Label, Single Site, 48 Week, Randomised Controlled Trial Evaluating the Safety and Efficacy of Exenatide Once-weekly in the Treatment of Patients With Multiple System Atrophy
Brief Title: Exenatide Once-weekly as a Treatment for Multiple System Atrophy
Acronym: MSA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 125591; 2020-000122-26 (EudraCT Number)
Record Dates: First submitted 2020-05-29; First posted 2020-06-16 (Actual); Results first posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Multiple System Atrophy
MeSH Terms: conditions — Multiple System Atrophy | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exenatide (Experimental)
  Interventions: Drug: Exenatide Pen Injector [Bydureon]
- Standard of care (No Intervention)

INTERVENTIONS:
Drug: Exenatide Pen Injector [Bydureon] — Exenatide is a treatment licensed for use in Type 2 diabetes.
  Arms: Exenatide

SUMMARY:
Fifty patients with early stage Multiple System Atrophy (MSA) will be recruited and randomised to receive Exenatide injections, or to act as controls in this open label trial. For half of the patients, Exenatide will be given as a once weekly subcutaneous injection in addition to participant's regular medication. All patients will continue to receive standard of care treatment for MSA. Detailed assessments will be made of all patients at baseline and periodically for a total of 48 weeks. The primary endpoint will be the difference in total Uniﬁed Multiple System Atrophy Rating Scale (UMSARS) score (Parts I and II) at 48 weeks comparing Exenatide treated to best medically treated patients (controls). Secondary measures will include adverse event reports, self-completed questionnaires, and blood test results. Aside from these assessments, all patients will continue any regular MSA medications throughout the trial with adjustments made only according to clinical need.

Standard of care treatment for patients on non IMP arm will be dependant on the patients individual symptoms - there is no broad standard treatment for every patient.

DETAILED DESCRIPTION:
Fifty patients with early stage MSA will be recruited and randomised to receive Exenatide injections, or to act as controls in this open label trial.

Once a potential participant has been identified they will receive a patient information leaflet, and will be given a minimum of 24 hours to read this before being recruited on to the trial. Patients will need to be eligible for the trial by meeting the inclusion criteria.

During pre-treatment there will be a screening visit and a baseline visit. Pre-treatment assessments will include: demographics, medical history, family history, any previous genetic tests recorded, previous drug compliance issues recorded, physical examination, neurological examination, 12-lead ECG, routine bloods (FBC, U&E, LFT, glucose, amylase, HbA1c, PT and APTT), height, weight, vital signs, serum or urine pregnancy tests (for women of childbearing potential), MoCA, BDI-II and Concomitant medications. Patients will then wear a sensor attached to their lower back for a week. They will then return for their baseline visit. At the baseline visit assessments will include: physical exam, neurological exam, lumbar puncture for CSF collection, serum collection, fasting blood tests, vital signs, UMSARS, COMPASS Select, COMPASS Change scale, timed motor tests, The Unified Dystonia Rating Scale, MoCA, BDI-II, Concomitant medication review and adverse event review. Participants will then be randomised to both control arm or trial drug arm and receive the according treatment. The baseline visit will also include a training session for self-administration of IMP.

Patients randomised to receive the trial drug will receive 2mg Exenatide once a week for 48 weeks via subcutaneous injection. Follow up visits will be every 12 weeks and patients will be given a sufficient supply to last them till their next follow up appointment (can be stored in fridge at home). They will also be given a dosing diary to record the time and day of injection administration.

Patients will continue to attend their normal neurology appointments as well as trial specific appointments. Patients will have a telephone call with the research nurse at week 4. Thereafter detailed assessments including Physical and Neurological exam, ECG's, Movement tests Including the Uniﬁed Multiple System Atrophy Rating Scale (videotaped), concomitant medications review, adverse event review, and blood sampling at baseline and every 12 weeks for a total of 48 weeks. Each patient will also have a Lumbar Puncture at baseline and at their final visit.

The primary endpoint will be the difference in total Uniﬁed Multiple System Atrophy Rating Scale (UMSARS) score (Parts I and II) at 48 weeks comparing Exenatide to best medically treated patients. Secondary measures will include adverse event reports, self-completed questionnaires, and blood test results. Aside from these assessments, all patients will continue any regular MSA medications throughout the trial with adjustments made only according to clinical need.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 30-80 years old with a diagnosis of Possible or Probable MSA of the parkinsonian subtype (MSA-P) or cerebellar subtype (MSA-C) according to The Gilman Criteria (Gilman et al. 2008).
* Participants who are less than five years from the time of documented MSA diagnosis or from the time of documented parkinsonian / ataxic neurological condition that later turns out to be MSA.
* Participants who are able to walk at least 10 metres with or without assistance. Participants with an anticipated survival of at least three years in the opinion of the investigator.
* Participants that are willing to adhere to the study drug regimen.
* Participants that are willing and able to perform all protocol-specified assessments and comply with the study visit schedule.
* Females of childbearing potential and male participants with partners of childbearing potential must agree to use an effective method of contraception from the time consent is signed until 10 weeks after treatment discontinuation. Females of childbearing potential have a negative pregnancy test within 7 days prior to being randomised.
* Willing and able to provide written informed consent.
* Subjects who are not able to write may give verbal consent in the presence of at least one witness, and the witness should sign the informed consent form.

Exclusion Criteria:

* Females who are pregnant, planning pregnancy or breastfeeding.
* Women of child-bearing potential who do not practice an acceptable method of birth control. Subjects who meet any of the following criteria which tend to suggest advance disease:

  1. Speech impairment as assessed by a score of ≥ 3 on UMSARS question 1
  2. Swallowing impairment as assessed by a score of ≥ 3 on UMSARS question 2
  3. Impairment in ambulation as assessed by a score of ≥ 3 on UMSARS question 7
  4. Falling more frequently than once per week as assessed by a score of ≥ 3 on UMSARS question 8. Participants with a clinically significant or unstable medical or surgical condition, which in the opinion of the investigator might preclude safe completion of the study.
* Participants with active malignant neoplasms or history of malignant neoplasm in the last 5 years. Participants with movement disorders other than MSA.
* Concurrent dementia defined by a score lower than 21 on the MoCA.
* Concurrent severe depression defined by a score of ≥30 on the Beck Depression Inventory-II.
* History of deep brain stimulation surgery.
* Participants who have taken any investigational products within 90 days prior to baseline.
* Participants with a BMI < 18.5.
* Participants with diabetes, end stage renal disease or severely impaired renal function.
* History of clinically significant cardiac disease, pancreatitis and/or alcoholism.
* Participants with severe gastrointestinal disease including gastroparesis.
* Ongoing treatment with sulphonylurea.
* Known allergies to the IMP and excipients of IMP.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Leonard Wolfson Experimental Neurology Centre, National Hospital of Neurology and Neurosurgery, UCLH NHS Foundation trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymised data will be made available from those patients who have provided consent to do so, following completion of trial data analysis, for any reasonable requests.

REFERENCES:
- [Background] Athauda D, Foltynie T. Insulin resistance and Parkinson's disease: A new target for disease modification? Prog Neurobiol. 2016 Oct-Nov;145-146:98-120. doi: 10.1016/j.pneurobio.2016.10.001. Epub 2016 Oct 3. PMID 27713036
- [Background] Athauda D, Foltynie T. The glucagon-like peptide 1 (GLP) receptor as a therapeutic target in Parkinson's disease: mechanisms of action. Drug Discov Today. 2016 May;21(5):802-18. doi: 10.1016/j.drudis.2016.01.013. Epub 2016 Feb 3. PMID 26851597
- [Background] Athauda D, Gulyani S, Karnati HK, Li Y, Tweedie D, Mustapic M, Chawla S, Chowdhury K, Skene SS, Greig NH, Kapogiannis D, Foltynie T. Utility of Neuronal-Derived Exosomes to Examine Molecular Mechanisms That Affect Motor Function in Patients With Parkinson Disease: A Secondary Analysis of the Exenatide-PD Trial. JAMA Neurol. 2019 Apr 1;76(4):420-429. doi: 10.1001/jamaneurol.2018.4304. PMID 30640362
- [Background] Athauda D, Maclagan K, Budnik N, Zampedri L, Hibbert S, Skene SS, Chowdhury K, Aviles-Olmos I, Limousin P, Foltynie T. What Effects Might Exenatide have on Non-Motor Symptoms in Parkinson's Disease: A Post Hoc Analysis. J Parkinsons Dis. 2018;8(2):247-258. doi: 10.3233/JPD-181329. PMID 29843254
- [Background] Athauda D, Maclagan K, Skene SS, Bajwa-Joseph M, Letchford D, Chowdhury K, Hibbert S, Budnik N, Zampedri L, Dickson J, Li Y, Aviles-Olmos I, Warner TT, Limousin P, Lees AJ, Greig NH, Tebbs S, Foltynie T. Exenatide once weekly versus placebo in Parkinson's disease: a randomised, double-blind, placebo-controlled trial. Lancet. 2017 Oct 7;390(10103):1664-1675. doi: 10.1016/S0140-6736(17)31585-4. Epub 2017 Aug 3. PMID 28781108
- [Background] Aviles-Olmos I, Dickson J, Kefalopoulou Z, Djamshidian A, Ell P, Soderlund T, Whitton P, Wyse R, Isaacs T, Lees A, Limousin P, Foltynie T. Exenatide and the treatment of patients with Parkinson's disease. J Clin Invest. 2013 Jun;123(6):2730-6. doi: 10.1172/JCI68295. PMID 23728174
- [Background] Aviles-Olmos I, Dickson J, Kefalopoulou Z, Djamshidian A, Kahan J, Ell P, Whitton P, Wyse R, Isaacs T, Lees A, Limousin P, Foltynie T. Motor and cognitive advantages persist 12 months after exenatide exposure in Parkinson's disease. J Parkinsons Dis. 2014;4(3):337-44. doi: 10.3233/JPD-140364. PMID 24662192
- [Background] Bassil, Fares, Marie-Hélène Canron, Anne Vital, Erwan Bezard, Pierre-Olivier Fernagut, and Wassilios G. Meissner. 2017. "Brain Insulin Resistance in Parkinson's Disease [MDS Abstracts]." Movement Disorders 32 (suppl.
- [Background] Bassil F, Canron MH, Vital A, Bezard E, Li Y, Greig NH, Gulyani S, Kapogiannis D, Fernagut PO, Meissner WG. Insulin resistance and exendin-4 treatment for multiple system atrophy. Brain. 2017 May 1;140(5):1420-1436. doi: 10.1093/brain/awx044. PMID 28334990
- [Background] Bergenstal RM, Wysham C, Macconell L, Malloy J, Walsh B, Yan P, Wilhelm K, Malone J, Porter LE; DURATION-2 Study Group. Efficacy and safety of exenatide once weekly versus sitagliptin or pioglitazone as an adjunct to metformin for treatment of type 2 diabetes (DURATION-2): a randomised trial. Lancet. 2010 Aug 7;376(9739):431-9. doi: 10.1016/S0140-6736(10)60590-9. Epub 2010 Jun 26. PMID 20580422
- [Background] Blevins T, Pullman J, Malloy J, Yan P, Taylor K, Schulteis C, Trautmann M, Porter L. DURATION-5: exenatide once weekly resulted in greater improvements in glycemic control compared with exenatide twice daily in patients with type 2 diabetes. J Clin Endocrinol Metab. 2011 May;96(5):1301-10. doi: 10.1210/jc.2010-2081. Epub 2011 Feb 9. PMID 21307137
- [Background] Consoli A, Formoso G. Potential side effects to GLP-1 agonists: understanding their safety and tolerability. Expert Opin Drug Saf. 2015 Feb;14(2):207-18. doi: 10.1517/14740338.2015.987122. Epub 2014 Dec 12. PMID 25496749
- [Background] Cork SC, Richards JE, Holt MK, Gribble FM, Reimann F, Trapp S. Distribution and characterisation of Glucagon-like peptide-1 receptor expressing cells in the mouse brain. Mol Metab. 2015 Aug 5;4(10):718-31. doi: 10.1016/j.molmet.2015.07.008. eCollection 2015 Oct. PMID 26500843
- [Background] D'Amelio M, Ragonese P, Callari G, Di Benedetto N, Palmeri B, Terruso V, Salemi G, Famoso G, Aridon P, Savettieri G. Diabetes preceding Parkinson's disease onset. A case-control study. Parkinsonism Relat Disord. 2009 Nov;15(9):660-4. doi: 10.1016/j.parkreldis.2009.02.013. Epub 2009 Apr 7. PMID 19356970
- [Background] Dodel R, Spottke A, Gerhard A, Reuss A, Reinecker S, Schimke N, Trenkwalder C, Sixel-Doring F, Herting B, Kamm C, Gasser T, Sawires M, Geser F, Kollensperger M, Seppi K, Kloss M, Krause M, Daniels C, Deuschl G, Bottger S, Naumann M, Lipp A, Gruber D, Kupsch A, Du Y, Turkheimer F, Brooks DJ, Klockgether T, Poewe W, Wenning G, Schade-Brittinger C, Oertel WH, Eggert K. Minocycline 1-year therapy in multiple-system-atrophy: effect on clinical symptoms and [(11)C] (R)-PK11195 PET (MEMSA-trial). Mov Disord. 2010 Jan 15;25(1):97-107. doi: 10.1002/mds.22732. PMID 20014118
- [Background] Drucker DJ, Buse JB, Taylor K, Kendall DM, Trautmann M, Zhuang D, Porter L; DURATION-1 Study Group. Exenatide once weekly versus twice daily for the treatment of type 2 diabetes: a randomised, open-label, non-inferiority study. Lancet. 2008 Oct 4;372(9645):1240-50. doi: 10.1016/S0140-6736(08)61206-4. Epub 2008 Sep 7. PMID 18782641
- [Background] Egan AG, Blind E, Dunder K, de Graeff PA, Hummer BT, Bourcier T, Rosebraugh C. Pancreatic safety of incretin-based drugs--FDA and EMA assessment. N Engl J Med. 2014 Feb 27;370(9):794-7. doi: 10.1056/NEJMp1314078. No abstract available. PMID 24571751
- [Background] Fanciulli A, Wenning GK. Multiple-system atrophy. N Engl J Med. 2015 Jan 15;372(3):249-63. doi: 10.1056/NEJMra1311488. No abstract available. PMID 25587949
- [Background] Fernagut PO, Dehay B, Maillard A, Bezard E, Perez P, Pavy-Le Traon A, Rascol O, Foubert-Samier A, Tison F, Meissner WG. Multiple system atrophy: a prototypical synucleinopathy for disease-modifying therapeutic strategies. Neurobiol Dis. 2014 Jul;67:133-9. doi: 10.1016/j.nbd.2014.03.021. Epub 2014 Apr 12. PMID 24727096
- [Background] Fineman MS, Mace KF, Diamant M, Darsow T, Cirincione BB, Booker Porter TK, Kinninger LA, Trautmann ME. Clinical relevance of anti-exenatide antibodies: safety, efficacy and cross-reactivity with long-term treatment. Diabetes Obes Metab. 2012 Jun;14(6):546-54. doi: 10.1111/j.1463-1326.2012.01561.x. Epub 2012 Feb 10. PMID 22236356
- [Background] Gilman S, Wenning GK, Low PA, Brooks DJ, Mathias CJ, Trojanowski JQ, Wood NW, Colosimo C, Durr A, Fowler CJ, Kaufmann H, Klockgether T, Lees A, Poewe W, Quinn N, Revesz T, Robertson D, Sandroni P, Seppi K, Vidailhet M. Second consensus statement on the diagnosis of multiple system atrophy. Neurology. 2008 Aug 26;71(9):670-6. doi: 10.1212/01.wnl.0000324625.00404.15. PMID 18725592
- [Background] Greig NH, Tweedie D, Rachmany L, Li Y, Rubovitch V, Schreiber S, Chiang YH, Hoffer BJ, Miller J, Lahiri DK, Sambamurti K, Becker RE, Pick CG. Incretin mimetics as pharmacologic tools to elucidate and as a new drug strategy to treat traumatic brain injury. Alzheimers Dement. 2014 Feb;10(1 Suppl):S62-75. doi: 10.1016/j.jalz.2013.12.011. PMID 24529527
- [Background] Low PA, Reich SG, Jankovic J, Shults CW, Stern MB, Novak P, Tanner CM, Gilman S, Marshall FJ, Wooten F, Racette B, Chelimsky T, Singer W, Sletten DM, Sandroni P, Mandrekar J. Natural history of multiple system atrophy in the USA: a prospective cohort study. Lancet Neurol. 2015 Jul;14(7):710-9. doi: 10.1016/S1474-4422(15)00058-7. Epub 2015 May 27. PMID 26025783
- [Background] Low PA, Robertson D, Gilman S, Kaufmann H, Singer W, Biaggioni I, Freeman R, Perlman S, Hauser RA, Cheshire W, Lessig S, Vernino S, Mandrekar J, Dupont WD, Chelimsky T, Galpern WR. Efficacy and safety of rifampicin for multiple system atrophy: a randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2014 Mar;13(3):268-75. doi: 10.1016/S1474-4422(13)70301-6. Epub 2014 Feb 5. PMID 24507091
- [Background] Madsbad S. Review of head-to-head comparisons of glucagon-like peptide-1 receptor agonists. Diabetes Obes Metab. 2016 Apr;18(4):317-32. doi: 10.1111/dom.12596. Epub 2015 Dec 29. PMID 26511102
- [Background] De Pablo-Fernandez E, Sierra-Hidalgo F, Benito-Leon J, Bermejo-Pareja F. Association between Parkinson's disease and diabetes: Data from NEDICES study. Acta Neurol Scand. 2017 Dec;136(6):732-736. doi: 10.1111/ane.12793. Epub 2017 Jun 26. PMID 28653373
- [Background] Poewe W, Hauser RA, Lang A; ADAGIO Investigators. Effects of rasagiline on the progression of nonmotor scores of the MDS-UPDRS. Mov Disord. 2015 Apr;30(4):589-92. doi: 10.1002/mds.26124. Epub 2014 Dec 27. PMID 25545629
- [Background] Poewe W, Seppi K, Fitzer-Attas CJ, Wenning GK, Gilman S, Low PA, Giladi N, Barone P, Sampaio C, Eyal E, Rascol O; Rasagiline-for-MSA investigators. Efficacy of rasagiline in patients with the parkinsonian variant of multiple system atrophy: a randomised, placebo-controlled trial. Lancet Neurol. 2015 Feb;14(2):145-52. doi: 10.1016/S1474-4422(14)70288-1. Epub 2014 Dec 8. PMID 25498732
- [Background] Talbot K, Wang HY, Kazi H, Han LY, Bakshi KP, Stucky A, Fuino RL, Kawaguchi KR, Samoyedny AJ, Wilson RS, Arvanitakis Z, Schneider JA, Wolf BA, Bennett DA, Trojanowski JQ, Arnold SE. Demonstrated brain insulin resistance in Alzheimer's disease patients is associated with IGF-1 resistance, IRS-1 dysregulation, and cognitive decline. J Clin Invest. 2012 Apr;122(4):1316-38. doi: 10.1172/JCI59903. PMID 22476197
- [Background] Wenning GK, Tison F, Seppi K, Sampaio C, Diem A, Yekhlef F, Ghorayeb I, Ory F, Galitzky M, Scaravilli T, Bozi M, Colosimo C, Gilman S, Shults CW, Quinn NP, Rascol O, Poewe W; Multiple System Atrophy Study Group. Development and validation of the Unified Multiple System Atrophy Rating Scale (UMSARS). Mov Disord. 2004 Dec;19(12):1391-402. doi: 10.1002/mds.20255. PMID 15452868
- [Background] Kollensperger M, Stampfer-Kountchev M, Seppi K, Geser F, Frick C, Del Sorbo F, Albanese A, Gurevich T, Giladi N, Djaldetti R, Schrag A, Low PA, Mathias CJ, Poewe W, Wenning GK. Progression of dysautonomia in multiple system atrophy: a prospective study of self-perceived impairment. Eur J Neurol. 2007 Jan;14(1):66-72. doi: 10.1111/j.1468-1331.2006.01554.x. PMID 17222116
- [Background] Wenning GK, Geser F, Krismer F, Seppi K, Duerr S, Boesch S, Kollensperger M, Goebel G, Pfeiffer KP, Barone P, Pellecchia MT, Quinn NP, Koukouni V, Fowler CJ, Schrag A, Mathias CJ, Giladi N, Gurevich T, Dupont E, Ostergaard K, Nilsson CF, Widner H, Oertel W, Eggert KM, Albanese A, del Sorbo F, Tolosa E, Cardozo A, Deuschl G, Hellriegel H, Klockgether T, Dodel R, Sampaio C, Coelho M, Djaldetti R, Melamed E, Gasser T, Kamm C, Meco G, Colosimo C, Rascol O, Meissner WG, Tison F, Poewe W; European Multiple System Atrophy Study Group. The natural history of multiple system atrophy: a prospective European cohort study. Lancet Neurol. 2013 Mar;12(3):264-74. doi: 10.1016/S1474-4422(12)70327-7. Epub 2013 Feb 5. PMID 23391524
- [Derived] Girges C, Vijiaratnam N, King A, Auld G, McComish R, Chowdhury K, Ambler G, Maclagan K, Limousin P, Athauda D, Morris HR, Libri V, Foltynie T; Exenatide PD3 and MSA Trials Consortia. Mild-to-moderate depressive symptoms impact on self-reported outcome measures in clinical trials for neurodegenerative diseases. Clin Trials. 2025 Nov 30:17407745251387571. doi: 10.1177/17407745251387571. Online ahead of print. PMID 41321006

RESULTS

PARTICIPANT FLOW:
Groups:
- Exenatide: Participants randomised to receive exenatide.
- Standard of Care: Participants randomised to receive standard care only.
Period: Overall Study
Arm/Group | Exenatide | Standard of Care
Started | 25 | 25
Completed | 21 | 23
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Death | 2 | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics includes all recruited participants, whereas the analysis only includes those who were followed-up for 48 weeks.
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide | Standard of Care | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: Age in years] | 63.3 (8.4) | 62.4 (7.3) | 63.3 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 12 | 12 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 25 | 50
  Unknown or Not Reported | 0 | 0 | 0
MSA Sub-type [Count of Participants; unit: Participants]
  MSA-P | 14 | 14 | 28
  MSA-C | 11 | 11 | 22
UMSARS (Part 1+2) [Mean (Standard Deviation); unit: Points] | 46.0 (11.1) | 42.6 (8.2) | 44.9 (9.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in UMSARS Score (Parts I+II) From Baseline
Description: The primary endpoint is the total Unified Multiple System Atrophy Rating Scale (UMSARS) score (Parts I and II), exploring the change from baseline overtime (evaluated at 48-weeks). Part I is a 12-item historical interview (max score 48) and Part II is a 14-item clinical examination (max score 56). Part I and II are added together to give a total score, which can range from 0 to 104. Higher scores indicate worse disease severity.
Time Frame: Baseline and 48 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Exenatide | Standard of Care
Number analyzed (Participants) | 24 | 24
score on a scale | 6.1 [3.0 to 9.3] | 13.3 [9.2 to 17.3]

2. Secondary Outcome: Loss of Independent Ambulation
Description: Proportion of participants with loss of independent ambulation, defined by a score of 4 on the UMSARS-I Item 7 (walking) at 48 weeks.
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide | Standard of Care
Number analyzed (Participants) | 25 | 25
Participants | 2 | 2

3. Secondary Outcome: Multiple System Atrophy Quality of Life (MSA-QoL) Scale
Description: The Multiple System Atrophy Quality of Life (MSA-QoL) scale measured health-related quality of life across three subscales (motor, nonmotor, and emotional/social functioning). Each item (40 in total) has five increasing levels of impairment (0 to 4), with 0 representing no impairment and 4 representing extreme impairment. Scores for the three subscales were generated by summing items and transformed to a range of 0 to 100 (100 × [(observed score minus min possible score)/(max possible score minus min possible score)]).
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Exenatide: Participants randomised to received exenatide.
Arm/Group | Exenatide | Standard of Care
Number analyzed (Participants) | 21 | 23
score on a scale
  MSA QoL (Motor Domain) | 53.1 (19.8) | 53.7 (23.7)
  MSA QoL (Non-motor Domain) | 37.4 (17.8) | 39.3 (15.4)
  MSA QoL (Emotional/Social Functioning Domain) | 33.3 (22.8) | 43.1 (23.9)

4. Secondary Outcome: Number of Falls
Description: Number of falls reported by the participant at 48-weeks.
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: Number of falls
Arm/Group | Exenatide | Standard of Care
Number analyzed (Participants) | 21 | 23
Number of falls | 1.7 (2.9) | 3.0 (6.8)

5. Secondary Outcome: Milestones on UMSARS Part 1 (Speech, Swallow and Falling)
Description: The UMSARS Part 1 is 12-item sub-scale which comprises a historic review of disease-related impairments. A single score using a 0 (no impairment) to 4 (severe impairment) was generated for each item (max score 48 points). We examined the proportion of participants reaching a score of ≥ 3 on UMSARS item 1 (speech), item 2 (swallowing) and item 8 (falling) by 48 weeks.
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide | Standard of Care
Number analyzed (Participants) | 21 | 23
Participants
  UMSARS Part 1 Item 1 (Speech) | 3 | 7
  UMSARS Part 1 Item 2 (Swallowing) | 2 | 8
  UMSARS Part 1 Item 8 (Falling) | 3 | 6

6. Secondary Outcome: Clinical Global Impression (CGI) Scale
Description: The CGI evaluates the change from the initiation of treatment on a seven-point scale (1 = =very much improved to 7 = very much worse since the initiation of treatment). A single score at 48 weeks was recorded.
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exenatide | Standard of Care
Number analyzed (Participants) | 21 | 23
score on a scale | 3.1 (1.0) | 2.4 (0.8)

7. Secondary Outcome: Montreal Cognitive Assessment (MoCA)
Description: The MoCA is a brief cognitive scale (scored out of 0-30 points). A score of 26 or more reflects normal cognitive abilities, whereas lower scores indicate cognitive impairment. The difference between groups (total score out of 30) was explored at 48 weeks.
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exenatide | Standard of Care
Number analyzed (Participants) | 21 | 23
score on a scale | 26.0 (2.7) | 27.2 (2.5)

8. Secondary Outcome: UMSARS Part IV
Description: The UMSARS Part 4 measures global disability (1 item) scored from 1 (completely independent) to 5 (totally dependent and helpless. Bedridden).
Time Frame: Score at 48 Weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Exenatide | Standard of Care
Number analyzed (Participants) | 21 | 23
Score on a scale | 2.8 (1.1) | 3.0 (0.9)

9. Secondary Outcome: Beck Depression Inventory II (BDI-II)
Description: The BDI-II is a self-report questionnaire designed to measure the severity of depression symptomatology (scored out of 0-63 points). A score of 13 or less indicated minimal, 14-19 indicated mild, 20-28 indicated moderate and 29-63 indicated severe depression. The difference between groups was explored at 48 weeks.
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Exenatide | Standard of Care
Number analyzed (Participants) | 21 | 23
Score on a scale | 14.3 (8.8) | 15.2 (8.0)

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Exenatide | Standard of Care
All-Cause Mortality (participants affected / at risk) | 2/25 | 2/25
Serious Adverse Events (participants affected / at risk) | 10/25 | 10/25
Other Adverse Events (participants affected / at risk) | 6/25 | 1/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide (N=25) | Standard of Care (N=25)
Anxiety (Psychiatric disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dysphagia (Nervous system disorders) | 0 | 4
Falls (Nervous system disorders) | 2 | 0
Hyponatremia (General disorders) | 0 | 1
Lung Infection (Infections and infestations) | 1 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sepsis (Infections and infestations) | 0 | 3
Serum Amylase Increased (Hepatobiliary disorders) | 2 | 0
Possible Detachment of Percutaneous Endoscopic Gastrostomy Tube (Surgical and medical procedures) | 0 | 1
Syncope (Cardiac disorders) | 2 | 0
Upper Respiratory Infection (Infections and infestations) | 3 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 0
Urinary Tract Infections (Infections and infestations) | 3 | 2
Vascular Disorders (Vascular disorders) | 0 | 1
Worsening of MSA (Nervous system disorders) | 2 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide (N=25) | Standard of Care (N=25)
Nausea (Gastrointestinal disorders) | 6 (9) | 1 (1) — Please see publication for full list of reported adverse events. We recorded total number of events per adverse event within each group, rather than recording how many participants were affected by each individual adverse event.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-06-13): https://cdn.clinicaltrials.gov/large-docs/13/NCT04431713/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/13/NCT04431713/SAP_001.pdf